CLINICAL TRIAL: NCT05822362
Title: Cannabidiol for Individuals at Risk for Alzheimer's Disease: A Randomized Placebo Controlled Trial
Brief Title: CBD for Individuals at Risk for Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-0619
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Cognition; Cannabidiol; Aging; Memory; Alzheimer's Disease; CBD; MCI; Mild Cognitive Impairment; Cognitive decline; Healthy aging; Older adults; Brain; Cannabis; Marijuana
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Marijuana Abuse | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: This is a double-blind, placebo-controlled, parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Full Spectrum Cannabidiol (Active Comparator): 200mg/day of full-spectrum cannabidiol, containing less than 0.3% THC.
  Interventions: Drug: Cannabidiol
- Broad Spectrum Cannabidiol (Active Comparator): 200mg/day of broad-spectrum cannabidiol, containing 0.0% THC.
  Interventions: Drug: Cannabidiol
- Hemp Seed Oil (Placebo Comparator): 200mg/day of hemp seed oil with no cannabinoids present.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cannabidiol — The current study will directly test the hypothesis that a moderate dose of CBD improves markers of Alzheimer's progression, cognitive function, sleep, pain, anxiety, oxidative stress, and inflammation.
  Other Names: CBD
  Arms: Broad Spectrum Cannabidiol; Full Spectrum Cannabidiol
Other: Placebo — Placebo arm.
  Arms: Hemp Seed Oil

SUMMARY:
This is a double-blind, randomized controlled trial designed to test the effects of cannabidiol (CBD) on validated biomarkers of Alzheimer's disease (AD) progression, and behavioral, neurocognitive, and clinical measures, with putative mechanisms of action.

DETAILED DESCRIPTION:
To better understand the effects of hemp-derived CBD with and without a small amount of THC, we propose a Phase II randomized clinical trial (RCT) to examine the clinical effects of Full Spectrum CBD (fsCBD, contains less than 0.3% THC) vs. Broad Spectrum CBD (bsCBD, does not contain THC), vs. a matching placebo in a population of individuals diagnosed with mild cognitive impairment (MCI).

This is a double-blind, placebo-controlled, parallel group study designed to assess the efficacy of fsCBD and bsCBD, compared to a placebo control, on biomarkers of Alzheimer's disease progression, cognitive function, pain, sleep quality, anxiety, oxidative stress, and inflammation. If eligible for the study, subjects will be randomized to receive one of the conditions for 24 weeks.

The current study will test the hypothesis that a moderate dose of CBD will improve measures of Alzheimer's disease progression, cognitive function, pain, sleep quality, anxiety, oxidative stress, and inflammation as compared to placebo. The study will also test whether endocannabinoids mediate the effects of CBD on these outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 55 - 85 and provide valid informed consent.
2. Participant must receive a diagnosis of Mild Cognitive Impairment after a careful cognitive and functional evaluation by a clinician.
3. Functional Activities Questionnaire (FAQ) score of 8 or less and self-reported ability to function independently
4. Montreal Cognitive Assessment (MoCa) score is between 18-25
5. Participant must have a CDR score of .5 on the Clinical Dementia Rating scale (CDR), which includes an assessment of function and is often used to distinguish MCI from dementia.
6. Must have an informant that will be utilized over the course of the 24 week study (must be the same person throughout study)
7. Participant must pass a test of consent comprehension
8. Must be interested in using CBD to help with cognitive function
9. Must plan on living in the Denver metro area over the next 6 months
10. Able to attend in-person visits at the study site

Exclusion Criteria:

1. Any other central nervous system (CNS) disease that would be expected to affect cognition, Parkinson's disease, multiple sclerosis.
2. Any history of brain injury (e.g., concussion with significant loss of consciousness)
3. Any significant systemic illness or unstable medical condition
4. Current use of Parkinson's medications, antipsychotic medications, anti-seizure medications, or anticholinergic medications
5. Current or lifetime diagnosis of a schizophrenia spectrum disorder, psychotic disorder, bipolar disorder type I & II, cluster B personality disorders (antisocial, borderline, narcissistic, histrionic), eating disorders, as defined by the DSM-5-TR
6. Participation in other clinical studies involving neuropsychological measures being collected more than one time per year.
7. Reported use of other drugs (cocaine, opiates, methamphetamine, MDMA) in the past 60 days or test positive on a urine test for those drugs of abuse at baseline.
8. Report using cannabis, including products with or without CBD, more than four times per month.
9. Recent history of, or meets criteria for major depression with suicidal ideation.
10. Reports use of medical CBD.
11. Liver function enzymes (AST, ALT) that are greater than 2x normal.
12. Currently taking medications known to be contraindicated with Epidiolex (buprenorphine, leflunomide, levomethadyl acetate, lomitapide, mipomersen, pexidartinib, propoxyphene, sodium oxybate, teriflunomide, clobazam, lamotrigine, valproate).
13. Pregnant at the time of study enrollment or unwilling to use contraception through the duration of the study (if not yet post-menopausal)
14. Individuals with potentially reversible causes of mild cognitive impairment (hypothyroidism, Vitamin B12 deficiency).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Function | Week 0 to Week 24
  The following assessments will be used to inform an aggregate measure of neurocognitive function:
  * The Clinical Dementia Rating Scale is a 5-point scale used to characterize six domains of cognitive and functional performance applicable to Alzheimer disease and related dementias. Higher scores indicate worse cognitive impairment.
  * NIH-Toolbox Cognitive Battery (NIH-TB CB) assessments are used to detect and measure specific aspects of cognition, including crystallized intelligence, psychomotor function, executive function, attention, and working memory.
  * Rey Auditory Verbal Learning Test to evaluate working memory and the Digit Symbol Substitution Task to evaluate global cognitive operations.
  * Montreal Cognitive Assessment (MoCa)
  * Functional Activities Questionnaire (FAQ) will be used to measure changes in dementia risk over the course of the clinical trial.
Biomarkers of Alzheimer's Disease Progression | Week 0 to Week 24
  * Changes in plasma levels of N-p-tau181 will be measured in ng/dl.
  * Changes in plasma Aβ42/Aβ40 ratio will be measured in ng/dl.
  * Changes in plasma Neurofilament Light (Nfl) will be measured in ng/dl.

SECONDARY OUTCOMES:
Change in pain | Week 0 to Week 24
  * The PROMIS Pain Intensity 1a questionnaire consists of two items asking about the participant's level of pain on average and at its worst in the past 7 days. Participants are asked to rate their pain on a scale from 0 (no pain) to 10 (worst imaginable pain).
  * The PROMIS Short Form v1.1 - Pain Interference - 6b scale will be used to assess how disruptive pain was over the past 7 days. There are six questions with a total score of 30-higher scores indicate more interference.
Change in sleep | Week 0 to Week 24
  * The PROMIS Sleep Disturbance 4a assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. Scores range from 4-20, with higher scores indicating worse sleep outcomes.
  * The PROMIS Sleep-Related Impairment 4a assesses perceptions of alertness, sleepiness, tiredness, and perceived functional impairments during usual waking hours due to sleep problems. Scores range from 4-20, with higher scores indicating worse sleep-related impairment.
  * The PROMIS Short Form v1.0 - Fatigue 4a measures subject fatigue over the past 7 days. Scores range from 4-20, with higher scores indicating more fatigue.
Change in anxiety | Week 0 to Week 24
  -The Depression Anxiety Stress Scale is a 21-item self-report instrument for measuring the three related negative emotional states of depression, anxiety, and tension/stress. Higher scores indicate worse anxiety
Change in plasma lipid biomarkers of inflammation and oxidative stress | Week 0 to Week 24
  Change in plasma levels of 5-iso PGF2αVI, 16-HETE, PGD2 will be measured in ng/dl.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado - Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No